CLINICAL TRIAL: NCT01898611
Title: Ghrelin Plus Strength Training in Frail Elderly Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anne Cappola, Division of Endocrinology, Diabetes, and Metabolism, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 818192
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Frailty Syndrome
Keywords: Frailty; Sarcopenia; Weight Loss; Exercise; Aging; Ghrelin; Elderly
MeSH Terms: conditions — Frailty; Sarcopenia; Weight Loss; Motor Activity | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ghrelin plus resistance training (Active Comparator): Ghrelin 7.5 mcg/kg as a once daily subcutaneous dose for 12 weeks plus resistance training
  Interventions: Drug: Ghrelin
- Placebo plus resistance training (Placebo Comparator): Placebo as a once daily subcutaneous dose for 12 weeks plus resistance training
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ghrelin — Ghrelin
  Arms: Ghrelin plus resistance training
Drug: Placebo — Saline will be used as a placebo
  Arms: Placebo plus resistance training

SUMMARY:
Frailty is a geriatric syndrome leading to physical deterioration including muscle wasting (sarcopenia) and unintentional weight loss. There are currently no approved therapies for frailty. Ghrelin is a hormone produced by the stomach that stimulates appetite centers in the brain. The investigators already know that a single dose of Ghrelin improves food intake immediately after the dose in frail older people. In addition, exercise programs have been shown to improve strength and function in older people. In this study, the investigators are trying to find out if a joint intervention of ghrelin and resistance training will improve walking, balance and leg strength in frail elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with three, four or five frailty criteria using the Fried frailty criteria

Exclusion Criteria:

1. Diabetes mellitus or fasting glucose ≥ 126 mg/dL
2. Hospitalization for stroke, myocardial infarction, coronary artery bypass graft surgery, vascular surgery in the past six months.
3. New York Heart Association Class III or IV congestive heart failure
4. Therapy for cancer in the past 12 months, except non-melanoma skin cancer
5. BMI ≥ 30 kg/m2
6. Current use of corticosteroids other than topical, ophthalmic, and inhaled preparations
7. Therapy with megestrol acetate or dronabinol within the last 6 weeks
8. Thyroid stimulating hormone measured as < 0.4 uIU/L or greater than 10uIU/L
9. Abnormal liver function tests (LFTs > 2x upper limit of normal)
10. Hemoglobin < 11g/dL
11. Insulin-like growth factor-I (IGF-I) above the age-specific reference range
12. History of surgery within the last 30 days
13. Hip fracture of hip or knee replacement within the previous 6 months or unable to walk
14. Deemed unsafe to participate by one of the study exercise therapists
15. Undergoing physical therapy or an exercise program
16. Unstable medical or psychological conditions or unstable home or food environment
17. Cognitive deficit as defined by a Folstein Mini Mental State Exam score < 24/30
18. Depression (defined as a score of > 11 on the Geriatric Depression Questionnaire)
19. Out of town for > 1 week during the 12 week study
20. Residing outside of a 15 mile radius of University of Pennsylvania Health System

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R. Cappola, M.D.,Sc.M., Principal Investigator — University of Pennsylvania, Perelman School of Medicine, Department of Medicine, Division of Endocrinology, Diabetes, and Metabolism
Locations (1):
- Clinical and Translational Research Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ghrelin Plus Resistance Training: Ghrelin 7.5 mcg/kg as a once daily subcutaneous dose for 12 weeks plus resistance training
  Ghrelin: 2:1 ratio placebo to ghrelin
  Resistance training: The exercise intervention will focus on twice weekly progressive strength training, taught by a certified fitness professional, to be performed in the home using dumbbells, an exercise step, and ankle weights.
- Placebo Plus Resistance Training: Placebo as a once daily subcutaneous dose for 12 weeks plus resistance training
  Resistance training: The exercise intervention will focus on twice weekly progressive strength training, taught by a certified fitness professional, to be performed in the home using dumbbells, an exercise step, and ankle weights.
Period: Overall Study
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Started | 5 | 11
Completed | 5 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.2 (4) | 81.6 (5) | 81.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Short Physical Performance Battery (SPPB)
Description: The SPPB includes three components: gait speed on a 15-foot walk, standing balance testing, and time to rise from a chair 5 times. Each test is rated on a five-level categorical score, with 0 representing inability to complete the test and 4 representing the highest level of performance, and summed to create a score ranging from 0 to 12.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
units on a scale | 0.6 (2.1) | 2.4 (1.7)

2. Primary Outcome: Treatment-associated Adverse Events
Description: Treatment-associated emergent adverse events, including clinically meaningful changes in laboratory measurements (IGF-1, HbA1c, fasting blood glucose, fasting insulin).
Time Frame: Twelve weeks
Measure: Number; unit: events
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
events | 0 | 0

3. Secondary Outcome: Change in Weight
Description: Change in weight from baseline to 12 weeks
Time Frame: Baseline to twelve weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
kg | -0.5 (0.5) | 0.88 (1.8)

4. Secondary Outcome: Change in Lean Body Mass
Description: Total lean body mass by dual energy x-ray absorptiometry
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
kg | 0.7 (0.8) | 1.0 (1.1)

5. Secondary Outcome: Change in Muscle Strength
Description: One repetition max bench press
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
kg | 16 (21) | 29 (25)

6. Secondary Outcome: Change in Food Intake
Description: Change in food intake by 3-day food intake record
Time Frame: Baseline to 12 weeks.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
kcal/day | 298 (127) | -81 (128)

7. Secondary Outcome: Change in Quality of Life
Description: Quality of life as assessed by short form 36 (SF-36), higher score indicates better quality of life, scale is 0-100 points
Time Frame: Baseline to 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
score on a scale | 8 (13) | 4 (8)

8. Secondary Outcome: Change in Frailty Status
Description: According to the Fried frailty criteria: Weight loss, exhaustion, low physical activity, slow walking speed, weakness, range 0 to 5, higher score indicates more frailty
Time Frame: Baseline to 12 weeks.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
Number analyzed (Participants) | 5 | 10
units on a scale | 3.2 [3 to 4] | 3.4 [3 to 4]

ADVERSE EVENTS:
Arm/Group | Ghrelin Plus Resistance Training | Placebo Plus Resistance Training
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/11
Other Adverse Events (participants affected / at risk) | 0/5 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ghrelin Plus Resistance Training (N=5) | Placebo Plus Resistance Training (N=11)
Pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No